CLINICAL TRIAL: NCT04026737
Title: Cardiovascular Effects of Chimeric Antigen Receptor T-Cell (CART Cell) Therapy: An Observational Prospective Study
Brief Title: Cardiovascular Effects of CART Cell Therapy
Acronym: CVE-CART
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC01419
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Leukemia; Lymphoma; Cardiotoxicity; Risk Factor, Cardiovascular; Immunotherapy
Keywords: Cardiotoxicity of Cancer Therapy; Cardio-Oncology; CART Cell Therapy
MeSH Terms: conditions — Leukemia; Lymphoma; Cardiotoxicity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — plasma, serum, and buffy are banked
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is an observational study aiming to prospectively define the rate of occurrence, natural history and progression of cardiac dysfunction in adults, and to identify the patients at high risk of developing cardiovascular events. The study enrolls patients prior to infusion with CART cell therapy and follows them with serial echocardiography, cardiac biomarkers, clinical data, and quality of life questionnaire.

DETAILED DESCRIPTION:
Patients have echo, blood draw, and QoL survey prior to CART infusion, then 2 days, 1 week, 1 month and 6 months following CART infusion. If patients experiences CRS, study team acquires echo within 72 hours of onset. As part of an optional substudy, patients wear an event monitor for 10 days, starting day of CART infusion.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Diagnosed with CD19+ malignancy undergoing treatment with CART cells

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with CD19+ malignancy (including but not limited to acute lymphoblastic leukemia, chronic lymphocytic leukemia, and difuse large B cell lymphoma) and scheduled for treatment with CART cells will be enrolled prior to infusion of CART cells.
Sampling Method: Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Left Ventricular (LV) Dysfunction | 6 months
  LV dysfunction, defined as a decrease in LV ejection fraction of at least 10% to less than or equal to 53%

SECONDARY OUTCOMES:
Incidence of Cardiovascular Events | 6 months
  Cardiovascular events are defined as hospitalization for symptomatic congestive heart disease, nonfatal acute coronary syndrome, cardiovascular death, nonfatal stroke, and all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Marielle Scherrer-Crosbie, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided